CLINICAL TRIAL: NCT06905717
Title: The T2D Profile - Studies of the Omics Profile in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: 448-16
Record Dates: First submitted 2021-03-02; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum, urine, feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The T2D Profile study examines the longitudinal molecular profiles of newly diagnosed type 2 diabetes (T2D), before and during guideline-based diabetes treatment.

DETAILED DESCRIPTION:
The study included a total of 3 visits: At baseline and after 1 and 3 months of diabetes treatment according to standard of care. Visits included clinical examinations, questionnaires and clinical chemistry. In addition, samples were collected at each visits for comprehensive molecular profiling including proteomics, genomics, transcriptomics, metabolomics, lipidomics, antibody profiling, mass cytometry and gene profiling of fecal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in the study.
* Age 50-65 years.
* T2D diagnosis (fasting p-glucose ≥7.0 mmol/L or an oral glucose tolerance test 2 hour p-glucose ≥11.1 mmol/L [or ≥12.2 mmol/L if measured capillary] at two separate occasions).

Exclusion Criteria:

* Diabetes medication before study start.
* Severe hyperglycemia requiring hospitalization or immediate insulin treatment, as judged by the investigator.
* Presence of any clinically significant disease which, in the opinion of the investigator, may interfere with the subject´s ability to participate in the study.
* Any major surgical procedure or trauma within 4 weeks of the first study visit.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with newly diagnosed Type 2 Diabetes identified from population-based cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Molecular profiles during diabetes treatment | 3 months
  Protein profiles will be compared between diabetes and control and diabetes treatment

CONTACTS AND LOCATIONS:
Overall Officials: Göran Bergström, MD, Prof, Principal Investigator — Göteborg University

REFERENCES:
- [Background] Gummesson A, Bjornson E, Fagerberg L, Zhong W, Tebani A, Edfors F, Schmidt C, Lundqvist A, Adiels M, Backhed F, Schwenk JM, Jansson PA, Uhlen M, Bergstrom G. Longitudinal plasma protein profiling of newly diagnosed type 2 diabetes. EBioMedicine. 2021 Jan;63:103147. doi: 10.1016/j.ebiom.2020.103147. Epub 2020 Dec 3. PMID 33279861